CLINICAL TRIAL: NCT00612989
Title: Phase I Trial of a 5-day Regimen of Temodar Plus O6-Benzylguanine (O6-BG) in the Treatment of Patients With Recurrent / Progressive Glioblastoma Multiforme
Brief Title: Ph I 5-day Temozolomide + O6-BG in Treatment of Pts w Recurrent / Progressive GBM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Schering-Plough (Industry); Keryx / AOI Pharmaceuticals, Inc. (Industry)
Responsible Party: David A. Reardon, MD, Duke University Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004058; 6788
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2009-01

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; GBM; Temodar; Temozolomide; O6-BG; O6-Benzylguanine; Recurrent GBM; Progressive GBM; Brain tumor; Malignant glioma; Neulasta; Pegfilgrastim
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Glioma | interventions — Temozolomide; O(6)-benzylguanine; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Schedule 1
  Interventions: Drug: Temodar and O6-Benzylguanine
- 2 (Experimental): Schedule 2
  Interventions: Drug: Temodar and O6-Benzylguanine
- 3 (Experimental): Schedule 2, Neulasta-supported
  Interventions: Drug: Temodar and O6-Benzylguanine

INTERVENTIONS:
Drug: Temodar and O6-Benzylguanine — O6-BG 120mg/m2 administered intravenously over 1 hr followed by continuous infusion of O6-BG at 30 mg/m2/day for 5 consecutive days. Every 48 hrs repeat dose of 120 mg/m2 over 1 hr administered for total of 3 doses.
  Temodar administered orally, in fasting state within 60 minutes of end of 1st 1-hr infusion of O6-BG & then every 24 hrs during continuous infusion of O6-BG. Temodar administered on day 1 of treatment cycle & every 24 hrs thereafter for 5 days with treatment cycles repeated every 28 days.
  Pts must fast for minimum of 1 hr prior to administration of each dose of Temodar & continue fasting 2 hrs after administration of each Temodar dose.
  Other Names: Temodar; Temozolomide; O6-BG; O6-Benzylguanine; NSC637037; Neulasta; Pegfilgrastim

SUMMARY:
Primary objectives To determine maxi tolerated dose of Temodar® in combo w O6-benzylguanine administered for 5 consecutive days in pts w progressive/recurrent GBM To characterize toxicity associated w Temodar® in combo w O6-BG administered for 5 consecutive days in pts w progressive/recurrent GBM To determine Neulasta®-supported MTD defined as the MTD of Temodar® in combo with O6-BG administered for 5 days while receiving Neulasta® once per treatment cycle between days 7 & 14 in pts w progressive/recurrent GBM To obtain preliminary response rates of Temodar® in combo w O6-BG administered for 5 consecutive days in pts w progressive/recurrent GBM

DETAILED DESCRIPTION:
1 primary objective is to determine maximum tolerated dose of Temodar in combo w O6-benzylguanine administered for 5 consecutive days in pts w progressive/recurrent GBM. Another primary objective is to characterize toxicity associated w Temozolomide in combo w O6-BG administered for 5 consecutive days in pts w progressive/recurrent GBM. 3rd primary objective is to determine Neulasta-supported MTD defined as MTD of Temozolomide in combo w O6-BG administered for 5 days while receiving Neulasta once per treatment cycle between days 7 & 14 in pts w progressive/recurrent GBM. Secondary objective is to obtain preliminary response rates of Temodar in combo w O6-BG administered for 5 consecutive days in pts w progressive/recurrent GBM. Population is Glioblastoma. O6-BG Administration: O6-BG 120mg/m2 administered intravenously over 1 hr followed by continuous infusion of O6-BG at 30mg/m2/day for 5 consecutive days. Every 48hrs repeat dose of 120mg/m2 over 1hr administered for total of 3 doses.

Temodar Administration: Temodar administered orally, in fasting state within 60 mins of end of 1st 1-hr infusion of O6-BG & then every 24 hrs during continuous infusion of O6-BG. Temozolomide administered on day 1 of treatment cycle and every 24 hrs thereafter for 5 days w treatment cycles repeated every 28 days. Body surface area calculated at beginning of each cycle will be used to calculate daily dose of Temozolomide administered for that cycle.

Neulasta Administration. Neulasta administered by subcutaneous injection in 0.6mL pre-filled syringe containing 6mg of pegfilgrastim. It will be administered once per chemotherapy cycle between days 7 & 14. Neulasta should not be administered in period between 14 days before & 24hrs after administration of cytotoxic chemo including Temozolomide.

Data Analysis will be conducted by Biostatistics department of Duke.

ELIGIBILITY:
Inclusion Criteria:

* Pts have histologically proven supratentorial GBM
* Pts have recurrent/progressive MG. If pt received stereotactic radiosurgery / brachytherapy as part of their prior therapy, then histologic confirmation of recurrence/metabolic imaging consistent w recurrent tumor is recommended but not mandated
* There must be measurable disease on contrast-enhanced magnetic resonance imaging study / CT scan performed <2wks of study drug administration
* Interval of >12 wks between completion of XRT & enrollment on protocol
* Interval of >4 wks between prior chemo & enrollment on protocol unless there is unequivocal evidence of tumor progression
* Interval of >2 wks between prior surgical resection & enrollment on protocol unless there is unequivocal evidence of tumor progression
* Age >18 yrs
* KPS >70 percent
* Following baseline study will be required <1wk of study drug administration: serum creatinine < 1.5 x ULN & Hematologic Status
* Following baseline studies will be required <1wk of study drug administration: absolute neutrophil count >2000 cells/microliter; platelet count >125,000 cells/microliter
* Following baseline studies will be required <1 wk of study drug administration: serum SGOT & total bilirubin < 2.5 x ULN
* Signed informed consent, approved by IRB, will be obtained prior to initiating treatment
* Pts w Reproductive Potential: Pts must agree to practice effective birth control measures while on study & for 2 months after completing therapy

Exclusion Criteria:

* Pregnant/breast feeding women/ women/men w reproductive potential not practicing adequate contraception. Therapy may be associated w potential toxicity to fetus/child that exceeds mini risks necessary to meet health needs of mother
* Prior treatment w O6-BG + Temozolomide in combo
* Active infection requiring intravenous antibiotics
* Known diagnosis of HIV infection
* Pts w history of another primary malignancy that is currently clinically significant/currently requires active intervention
* Pts unwilling/unable to comply w protocol due to serious medical/psychiatric condition
* Pts who have received investigational drugs <2 wks prior to start on study drug/have not recovered from side effects of such therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2005-02; Primary Completion 2007-08 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 6 months

SECONDARY OUTCOMES:
Progression-free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/